CLINICAL TRIAL: NCT00363259
Title: Pegintron Induction Therapy in Previous Non-Responders With Chronic HCV: A Dutch Multicenter Randomized Controlled Trial. (PIT-Study)
Brief Title: Pegintron Induction Therapy in HCV Non-Responders
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Foundation for Liver Research (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCV01-01
Record Dates: First submitted 2006-08-10; First posted 2006-08-15 (Estimated); Last update posted 2006-08-15 (Estimated); Status verified 2006-08

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — peginterferon alfa-2b; Ribavirin

INTERVENTIONS:
Drug: Peginterferon alfa-2b
Drug: Ribavirin

SUMMARY:
The purpose of this study is to compare the sustained virological response rate at 24 weeks after the end of experimental treatment (induction and 72 weeks) to that of standard 48 weeks treatment with PEG-inteferon alfa-2b and ribavirin in patients with chronic hepatitis C previous unresponsive to interferon alfa monotherapy or interferon alfa/ribavirin combination therapy.

ELIGIBILITY:
Inclusion Criteria:

* chronic hepatitis C
* non-response or relapse to previous interferon therapy with or without ribavirin for at least 3 months at any previous time
* detectable serum HCV-RNA
* elevated serum ALT activity documented on at least two occasions within the past 12 months, with at least one during the 90 day screening period preceding the initiation of test drug dosing
* liver biopsy findings (during screening or within previous 12 months) consistent with active fibrosis (haemophiliacs are excluded from biopsies)
* compensated liver disease (Child-Pugh Grade A clinical classification)
* negative urine or blood pregnancy test (for women of childbearing potential) documented within the 24-hour period prior to the first dose of study drug
* all fertile males and females receiving ribavirin and their fertile or potentially fertile partners must be advised to use two forms of effective contraception (combined) during treatment and during the 6 months after end of treatment

Exclusion Criteria:

* history or other evidence of severe illness, malignancy or any other condition which would make the patient, in the opinion of the investigator, unsuitable for the study
* women with ongoing pregnancy or breast feeding
* therapy with any systemic anti-viral, anti-neoplastic or immunomodulatory treatment (including supraphysiologic doses of steroids and radiation) <3 months prior to the first dose of study drug
* any investigational drug <6 weeks prior to the first dose of study drug
* positive test at screening for HBsAg, anti-HIV Ab
* history or other evidence of bleeding from esophageal varices, ascites, or other conditions consistent with decompensated liver disease (Child-Pugh Grade B or C clinical classification)
* Signs or symptoms of hepatocellular carcinoma
* history or other strong evidence of a medical condition associated with chronic liver disease other than HCV (e.g., primary hemochromatosis, autoimmune hepatitis, metabolic liver disease, alcoholic liver disease, toxin exposures
* Hb <7.5 mmol/l in women or <8.6 mmol/l in men at screening
* any patient with an increased baseline risk for anaemia (e.g. thalassemia, spherocytosis, etc) or for whom anaemia would be medically problematic
* neutrophil count <1500 cells/mm3 or platelet count <80,000 cells/mm3 at screening
* serum creatinine level >1.5 times the upper limit of normal at screening
* history of severe psychiatric disease, especially depression
* history of a severe seizure disorder or current anticonvulsant use
* history of immunologically mediated disease
* history or other evidence of chronic pulmonary disease associated with functional limitation
* history of severe allergies
* history of symptomatic and/or significant cardiovascular disease
* poorly controlled diabetes mellitus
* history of major organ transplantation with an existing functional graft
* hyper- or hypothyroidism
* evidence of severe retinopathy
* evidence of drug abuse (including excessive alcohol consumption within one year before study entry

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110
Dates: Start 2002-07; Study Completion 2005-11

PRIMARY OUTCOMES:
sustained virological response (HCV-RNA negative 24 weeks after end of treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Rob J de Knegt, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (7):
- Netherlands (7):
  - OLVG, Amsterdam
  - Rijnstate Ziekenhuis, Arnhem
  - Atrium Medisch Centrum, Heerlen
  - LUMC, Leiden
  - Erasmus MC, Rotterdam
  - Ziekenhuis Zeeuws Vlaanderen, Terneuzen
  - UMC, Utrecht